CLINICAL TRIAL: NCT06261411
Title: Effects of Replacing Routine Chest Radiography With Lung Ultrasound for Patients Undergoing Thoracic Surgery: A Randomised Controlled Trial
Brief Title: Lung Ultrasound as Alternative to Radiography in Thoracic Surgery
Acronym: LUS-ART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Sebastian Ullmark, Principal Investigator, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 999430; FOU2024-00038 (Registry Identifier: Forskning och Utveckling (Region Uppsala))
Record Dates: First submitted 2024-01-30; First posted 2024-02-15 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Thoracic Surgery; Ultrasonography
Keywords: Thoracic surgery; Lung ultrasound; Chest X-ray; Nurse

STUDY DESIGN:
Intervention Model Description: Case-Control
Who Masked: Outcomes Assessor
Masking Description: Inter-rater variability will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung Ultrasound (Experimental): Lung ultrasound based on specified protocol as primary method of investigation
  Interventions: Diagnostic Test: Lung Ultrasound
- Routine Care (No Intervention): Routine care defined as conventional chest x-ray as primary method of investigation

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound — Diagnostic ultrasound of pulmonary tissues such as pleura, plural spaces, and parenchyma.
  Other Names: LUS
  Arms: Lung Ultrasound

SUMMARY:
This projects aim is to study the effects of substitute conventional chest x-ray with lung ultrasound for patients undergoing thoracic surgery.

Participants in the study will be randomized to either ultrasound or routine chest x-ray as the primary method of diagnosis after having received surgery to their lungs.

DETAILED DESCRIPTION:
Modern lung surgery involves a variety of procedures that expose patients to the risk of developing postoperative complications (PPC). In lung surgery such as resections or lobectomies where a part of the lung tissue is removed, so-called single-lung ventilation is used. Through this technique, the lung that is operated on collapses, while ventilation is directed to the lung that is not operated on. When the operation is over, the structures of the lung are sewn together and the collapsed lung is inflated again. At this stage, it is important to ensure that the expansion of the lung is adequate. It is also important for the continued expansion of the lung that there is no air leakage from the lung to the pleural cavity. Therefore, there is initially a drainage in the pleural cavity to prevent both bleeding and air leakage. Postoperatively, several X-ray examinations are performed before the patient is discharged to ensure adequate lung expansion.

Lung ultrasound is a well-established method that is based on physical artifacts that arise in the interaction between ultrasound and various conditions in the lung tissue. The method is used in most of the questions that are usually asked even in chest X-rays and other conventional techniques but has the advantages of being both cost- and time-effective and does not involve the radiation dose that conventional X-rays involve.

The study aims to investigate whether lung ultrasound can replace conventional chest X-rays in patients who have undergone lung surgery. The research subjects will be randomized to undergo postoperative lung ultrasound or conventional chest X-rays after lung surgery.

Previous research has shown the possibility of abandoning X-ray radiation in favor of ultrasound in most scenarios. However, randomized studies are generally lacking, especially in this population.

ELIGIBILITY:
Inclusion Criteria:

* Segmental, partial, or wedge resection lung surgery, or lobectomy.
* Written informed consent
* Available research team for measurements.

Exclusion Criteria:

* Pregnancy
* Re-surgery due to complications related to the original surgery
* Need for critical care or admittance to the ICU.
* Patient or physician choice of withdrawal from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in chest x-ray | Through patient hospital stay, an average of five days
  Reduction in chest x-ray in patients undergoing thoracic surgery when LUS is the primary method of investigation.

SECONDARY OUTCOMES:
Re-insertion of chest tube | Through patient hospital stay, an average of five days
  The need for re-insertion och chest tube because of clinical deterioration, and/or verified clinically relevant post-operative pulmonary complication
Delayed removal of chest tube | Through patient hospital stay, an average of five days
  Number of patients in need of prolonged care with chest tube.
Time to chest tube removal | Through patient hospital stay, an average of five days
  Time, in hours, to eventual removal of chest tube
Patient Satisfaction | Through patient hospital stay, an average of five days
  Sub-group analysis of the patient experience and satisfaction for patients receiving both lung ultrasound and chest x-ray, measures through quantitative psychometric questionnaire with Likert-design consisting of a minimum value of 1 and a maximum of 5. Worse outcome is associated with low scores and vice versa.

OTHER OUTCOMES:
Missed Care | Through patient hospital stay, an average of five days
  The number of missed diagnoses of post-operative pulmonary complications based on results from chest x-ray in patients subjected to group crossover.
Inter-rater variability | Through patient hospital stay, an average of five days
  Inter-observer agreement study of collected ultrasound images.

CONTACTS AND LOCATIONS:
Overall Officials: Laila Hellgren-Johansson, PhD, Study Director — Region Uppsala
Locations (1):
- Uppsala Akademiska sjukhuset, Uppsala, Uppland, Sweden

DOCUMENTS (3):
  • Study Protocol (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT06261411/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT06261411/SAP_002.pdf
  • Informed Consent Form (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT06261411/ICF_001.pdf